CLINICAL TRIAL: NCT05657938
Title: A Phase 0 Study to Evaluate the Clinical Readiness of a Wearable Sensor Device and Duchenne Video Assessment in the Home Environment on Participants With Duchenne Muscular Dystrophy (DMD)
Brief Title: Evaluation of Home Based Assessments on Participants With DMD
Status: Completed | Type: Observational
Sponsor: Solid Biosciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SB-000-22-001
Record Dates: First submitted 2022-10-26; First posted 2022-12-20 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: duchenne; muscular dystrophy; DMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies | interventions — Wearable Electronic Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DMD Patients: Ambulatory males aged 4 to <13 years with Duchenne Muscular Dystrophy
  Interventions: Device: Wearable Device; Other: Duchenne Video Assessment (DVA)
- Age Matched Controls: Normal male age-matched controls
  Interventions: Device: Wearable Device; Other: Duchenne Video Assessment (DVA)

INTERVENTIONS:
Device: Wearable Device — The wearable device used in this study is an FDA 510(k) cleared Class II medical device designed to collect medical grade, clinical quality biometric, physiological and other electronic clinician outcome assessments data in a clinical trial setting. The system processes raw data into recognizable clinical metrics including vital signs, activity and posture classifications, surface electromyography (sEMG), and sleep metrics. The sensors are multi-modal, multilocation, rechargeable and reusable.
Other: Duchenne Video Assessment (DVA) — The DVA is a standardized tool that documents and assesses compensatory movement strategies as a marker of quality of movement.

SUMMARY:
This study is designed to evaluate the feasibility, wearability and participant satisfaction of novel outcome assessment tools in DMD patients which are performed in the home environment.

DETAILED DESCRIPTION:
This is a low interventional feasibility study to evaluate the use of:

1. An FDA 510(k) cleared Class II wearable medical device designed to collect medical grade, clinical quality biometric, physiological and other electronic clinician outcome assessments data in a clinical trial setting, and;
2. The Duchenne Video Assessment (DVA) tool to evaluate the quality of movement in patients with Duchenne Muscular Dystrophy (DMD)

This study will provide data on suitability of these tools in future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

For DMD patients:

1. Parent/guardian or participant is able to give informed consent and/or assent as required by local regulations, and all are willing and able to comply with the protocol.
2. Participant is assigned male sex at birth and is age 4 to <13 years at time of consent.
3. Participant has a confirmed diagnosis of DMD based on genetic testing and/or clinical records consistent with the diagnosis.
4. Participant has been on a stable glucocorticoid dose for 3 months prior to participation.
5. Participant is ambulatory as defined by the ability to walk down a hallway at home without assistance or support.

For healthy age-matched controls:

1. Parent/guardian or participant is able to give informed consent and/or assent as required by local regulations, and all are willing and able to comply with the protocol.
2. Participant is assigned male sex at birth and age 4 to <13 years at time of consent.

Exclusion Criteria:

For DMD Patients:

1. Participant is/was enrolled in any interventional study for DMD in the past 3 months or has ever been enrolled in a gene therapy study.
2. Participant is on any approved therapy for DMD except for glucocorticoids.
3. Participant is currently or was previously treated with exon-skipping antisense oligonucleotides such as eteplirsen, golodirsen, casimersen, and viltolarsen.
4. Participant has any prior or ongoing medical condition, medical history, or physical finding that could affect the participant's ability to perform the study assessments.
5. Participant has had major surgery within 3 months prior to recruitment or planned orthopedic surgery for any time during this study which would interfere with the ability to perform assessments.
6. Participant has a history of allergic response to silicones or adhesives.
7. Participant has an active implanted device (e.g., pacemaker). Implanted devices relying on an electrical power source to function are considered active devices.

For healthy age-matched controls:

1. Participant has a known musculoskeletal disease or had a musculoskeletal injury in the past 3 months.
2. Participant has other illness that precludes functional testing.
3. Participant is enrolled in any interventional study.
4. Participant has or has had any prior or ongoing medical condition, medical history, or physical finding that could affect the participant's ability to perform the study assessments.
5. Participant has had major surgery within 3 months prior to recruitment or planned orthopedic surgery for any time during this study which would interfere with the ability to perform study assessments.
6. Participant has a history of allergic response to silicones or adhesives.
7. Participant has an active implanted device (e.g., pacemaker). Implanted devices relying on an electrical power source to function are considered active devices.

Ages: 4 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Study Population: Approximately twenty ambulatory males aged 4 to <13 years with DMD will be recruited. Of these, approximately 10 participants will be considered Early Ambulatory and 10 will be considered Late Ambulatory. Early ambulatory is defined as able to get off the floor without assistance or use of furniture.
  Approximately twenty healthy, age-matched controls will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Wearable sensor device compliance | 30 days
  The wearable sensor device is composed of three small sticker-based sensors that are worn on the chest, thigh and ankle to record activity. Participants will wear the sensors during specified periods over the study duration and compliance will be assessed based on recorded activity.
Accuracy of functional evaluation using the Duchenne Video Assessment (DVA) tool in an at-home setting | 30 days
  The DVA is a digital tool designed to remotely evaluate functional capacity in a natural environment. Participants will complete a set of movement tasks at specified timepoints during the study that will be captured on video and scored by remote evaluators. DVA scoring will be compared with anticipated levels of functional capacity to assess accuracy.
Preference for use of the wearable sensor device and DVA tool as assessed by interview | Day 24-30
  Participants will be asked to complete an exit interview at the conclusion of the study to assess user preference.

CONTACTS AND LOCATIONS:
Overall Officials: Carl A Morris, PhD, Study Director — Solid Biosciences
Locations (1):
- Solid Biosciences, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No